CLINICAL TRIAL: NCT00289562
Title: A Phase I/II, Multi-Center, Open-Label, Repeat-Dose Study of Forodesine Hydrochloride Infusion in Patients With B-Cell Acute Lymphoblastic Leukemia With an Option of Extended Use of Forodesine Hydrochloride
Brief Title: Forodesine Hydrochloride (BCX-1777) for B-Cell Acute Lymphoblastic Leukemia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: BioCryst Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BCX1777-Bi-04-106
Record Dates: First submitted 2006-02-08; First posted 2006-02-10 (Estimated); Last update posted 2012-01-20 (Estimated); Status verified 2012-01

CONDITIONS: B-cell Acute Lymphoblastic Leukemia
Keywords: B-cell; leukemia; B-lymphoblastic leukemia; lymphoma; B-All
MeSH Terms: conditions — Burkitt Lymphoma; Leukemia; Lymphoma | interventions — forodesine

INTERVENTIONS:
Drug: forodesine hydrochloride (BCX-1777)

SUMMARY:
A Phase I/II, Multi-Center, Open-Label, Repeat-Dose Study of Forodesine Hydrochloride Infusion in Patients with B-cell Acute Lymphoblastic Leukemia with an Option of Extended Use of Forodesine Hydrochloride

ELIGIBILITY:
Inclusion Criteria:

* Documented B-cell acute lymphoblastic leukemia (B-ALL), which under WHO Guidelines is now referred to as precursor B-lymphoblastic leukemia/lymphoma
* Must have failed at least 1 treatment regimen for B-ALL, which under WHO Guidelines is now referred to as precursor B-lymphoblastic leukemia/lymphoma
* Performance status of ≤2 by Eastern Cooperative Oncology Group (ECOG) criteria
* Any age is allowed
* Life expectancy of at least 3 months
* Adequate liver function (aspartate transaminase [AST] and/or alanine transaminase [ALT] not >3 times upper limits of normal [ULN])
* Adequate kidney function (calculated creatinine clearance >40 mL/min)
* Negative serum or urine pregnancy test within 2 to 7 days prior to the start of study treatment in females of childbearing potential
* Females of childbearing potential and males must be willing and able to use an adequate method of contraception to avoid pregnancy for the duration of the study in such a manner that the risk of pregnancy is minimized. Acceptable contraceptives include intra-uterine devices (IUDs), hormonal contraceptives (oral, depot, patch, or injectable) and double barrier methods such as condoms or diaphragms with spermicidal gel or foam.
* Signed informed consent form (ICF), minor assent form (if applicable), prior to start of any study-specific procedures

Exclusion Criteria:

* Active serious infection not controlled by oral or intravenous antibiotics
* Treatment with any investigational antileukemic agent or chemotherapy agent in the last 7 days prior to study entry and lack of full recovery from side effects due to prior therapy independent of when that therapy was given
* Rapidly progressive disease with compromised organ function judged to be life-threatening by the Investigator
* Patients with clinical evidence of active central nervous system (CNS) disease
* Concurrent treatment with other anticancer agents
* Pregnant and/or lactating female
* Patients with known human immunodeficiency virus (HIV) infection HIV testing will be performed at the Screening visit for patients who have not been tested within 6 months of receiving study drug, as well as those patients who have had exposure or have been transfused with blood products that were not appropriately screened.
* Patients with known active hepatitis B and/or hepatitis C infection Hepatitis testing will be performed at the Screening visit for patients who have not been tested within 6 months of receiving study drug, as well as those patients who have had exposure or have been transfused with blood products that were not appropriately screened.
* Hypersensitive or intolerant to any component of the study drug formulation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20
Dates: Start 2004-09; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Denver, Colorado
  - Chicago, Illinois
  - Kansas City, Kansas
  - New York, New York
  - Houston, Texas
  - Abingdon, Virginia